CLINICAL TRIAL: NCT03169257
Title: Paediatric Obesity and Cardiovascular Dysfunction: Searching for Early Markers of Damage
Brief Title: Paediatric Obesity and Cardiovascular Dysfunction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Azienda Ospedaliero Universitaria Maggiore della Carita (Other)
Responsible Party: Principal Investigator, Flavia Prodam, Associated professor, Azienda Ospedaliero Universitaria Maggiore della Carita
Allocation: Non-Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: CE 95/12
Record Dates: First submitted 2017-05-24; First posted 2017-05-30 (Actual); Last update posted 2023-07-24 (Actual); Status verified 2020-07

CONDITIONS: Obesity, Childhood; Cardiovascular Diseases
Keywords: paediatric obesity; cardiovascular dysfunction; metabolic syndrome; adipokines; inflammation; oxidative stress
MeSH Terms: conditions — Pediatric Obesity; Cardiovascular Diseases; Metabolic Syndrome; Inflammation | interventions — Diet; Exercise

STUDY DESIGN:
Intervention Model Description: Only one group, the obese children group (OB) will be followed for one year. At baseline they received a behavioral intervention which comprises a Mediterranean balanced diet plus daily aerobic training.
Who Masked: Outcomes Assessor
Masking Description: A sonographer will perform cardiovascular imaging. Images will be reviewed by an expert pediatric cardiologist and an expert vascular surgeon blinded to patients' clinical data.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- OB (Experimental): Obese subjects according to the International Obesity Task Force (IOTF) criteria aged 6 to 16 years. OB subjects will undergo for 12 months an isocaloric Mediterranen balanced diet plus a daily aerobic training for at least 60 minutes.
  Interventions: Behavioral: diet plus physical activity
- NW (No Intervention): Normal weight subjects according to the International Obesity Task Force (IOTF) criteria aged 6 to 16 years and age, sex and pubertal status matched with the OB group

INTERVENTIONS:
Behavioral: diet plus physical activity — OB subjects will undergo an isocaloric Mediterranen balanced diet plus a daily aerobic training for at least 60 minutes. All the evaluations will be performed at baseline and after 6 and 12 months of this behavioral therapy. To assess food consumption, foods will be divided according to the classic basic food groups by the Italian Institute of Research on Food and Nutrition. Food frequencies questionnaires, validated for a wide range of ages, will be also completed by parents. Physical activity will be recorded by parents daily on a specific questionnaire.
  Arms: OB

SUMMARY:
Background Childhood obesity has been related to an impaired cardiovascular structure and function. Aims of this study will be to evaluate early cardiovascular abnormalities in a large population of obese children and adolescents compared with a normal weight counterpart, to investigate the potential association with insulin resistance (IR), serum uric acid (sUA), metabolic syndrome (MetS), plasmatic markers of inflammation and oxidative stress and adipokines, to evaluate changes in cardiovascular dysfunction after 6 and 12 months of a behavioral treatment (isocaloric Mediterranean balanced diet plus daily aerobic physical activity).

Subjects and methods This was a single-center case-control study. Eighty obese (OB) subjects (6-16 years) and 20 normal weight (NW) matched controls were consecutively recruited. In the whole population we will perform an anthropometric and a cardiovascular assessment. OB patients will also undergo an OGTT and biochemical evaluations. In the OB group, all these evaluations will be performed at baseline and after 6 (T6) and 12 months (T12) of diet plus aerobic training.

DETAILED DESCRIPTION:
Background Childhood obesity causes a wide range of severe complications, increasing the risk of premature morbidity and mortality and raising public-health concerns. In addition, obese children are more prone to become obese adults, with higher risk of cardiovascular diseases (CVD). A cluster of CVD risk factors has been identified in children as young as 5 years of age. Furthermore, among adolescents and young adults, the presence of CVD risk factors correlates with asymptomatic coronary atherosclerosis. Childhood obesity has been related to an impaired cardiac structure and function.

Atherogenesis and arterial wall damage begin during childhood and, there is evolving evidence that clinical indicators of atherosclerosis such as carotid artery intima-media thickness (CIMT), arterial stiffness, and endothelial function are altered in obese children. In addition, little is known on the potential association between early cardiovascular alterations and metabolic abnormalities in obese children. Metabolic syndrome (MetS) is a cluster of features, which includes dyslipidemia, hypertension, and visceral obesity, conferring with a higher risk of CVD and type 2 diabetes. Few studies investigated the association of MetS with cardiovascular changes during childhood. Hyperuricemia has been recognized as a risk factor for CVD in adults with a negative impact on longevity. However, data in pediatric age are still lacking and the association between hyperuricaemia and cardiovascular abnormalities in obese children is still unknown. Furthermore, obesity is a state of chronic low-level inflammation and increased oxidative stress. Oxidative stress plays an important role in the pathogenesis of cardiovascular alterations by either triggering or exacerbating the biochemical processes accompanying endothelial dysfunction.

Moreover, adipose tissue acts as a secretory gland, releasing hormones and adipokines with pro- or anti-inflammatory activity. Clinical studies of obese adults have observed an association between plasma levels of adipokines and markers of inflammation and/or oxidative stress. Among various adipokines, adiponectin seems to play an important role. Indeed, in contrast to other adipokines which are up-regulated in obesity, secretion of adiponectin is markedly reduced in obese subjects. Second, adiponectin seems to exert mainly positive activities on metabolism, vascular tone and inflammatory reaction. Consequently, in contrast to other adipokines, which circulate in excess in obese subjects and exert unbeneficial effects when chronically elevated, deficiency rather than excess of adiponectin is implicated in obesity-associated complications. Finally, serum concentration of adiponectin is very high in comparison to other hormones and cytokines, which suggests that apart from binding to specific high-affinity receptors, this protein may also have some less specific low affinity targets. Adiponectin has been associated with endothelial improvement and vascular protection through the activation of an endothelial isoform of nitric oxide (eNOS)-related signalling and with anti-inflammatory properties and antiatherogenic effects. Thus, an impaired production of adipokines may be a key mechanism linking obesity with inflammation and oxidative stress. The understanding of these complex mechanisms and the identification of possible early markers of cardiovascular damage are therefore necessary in order to establish preventive and therapeutic measures in childhood and to decrease cardiovascular morbidity and mortality in adulthood.

Subjects and methods This study is a single-centre longitudinal study. Subjects were recruited at Division of Pediatrics, Department of Health Sciences, University of Piedmont Orientale, Novara (Italy). The study protocol was in accordance with the ethical guidelines of the Declaration of Helsinki and has been approved by the local Ethical Committee. Informed written consent was obtained from all subjects and their parents before study. The investigators consecutively enrolled 80 Caucasian obese (OB) children and adolescents, aged 6 to 16 years, and 20 normal weight, age and sex matched controls (NW). NW patients were evaluated only at baseline while OB subjects will be evaluated at baseline and after 6 (T6) and 12 months (T12) of an isocaloric Mediterranean balanced diet plus aerobic training.

Assessment in both groups (OB and NW)

Echocardiographic assessment Transthoracic echocardiogram using a Vivid 7 Pro ultrasound scanner (General Electric Healthcare, USA) will be performed by a sonographer and the images will be reviewed by an expert pediatric cardiologist, blinded to patients' clinical data. Measurements of left ventricle (LV end-diastolic diameter, LVEDD; LV end-systolic diameter, LVESD; interventricular septum at end diastole, IVSD; LV posterior wall at end diastole, LVPWD) and left atrium diameter (LAD) will be obtained according to established standards. The maximum LA volume will be calculated from apical 4- and 2-chamber zoomed views of the LA. LV end-diastolic and end-systolic volumes and the LV ejection fraction at rest will be computed from 2- and 4-chamber views, using a modified Simpson's biplane method. LV mass (LVM) will be derived from the Devereux formula and indexed to body surface area (left ventricular mass index [LVMI]). Relative wall thickness (RWT) will be calculated as the ratio (LVPWD x 2)/LVEDD. Using pulsed wave Doppler, mitral inflow velocities, peak early diastolic velocity (E), peak late diastolic velocity (A), E/A ratio, will be measured.

Vascular assessment Vascular measurements will be performed with a high-resolution ultrasonography (Esaote MyLab25TM Gold, Esaote, Italy) using a 8-megaHertz (mHz) linear transducer and a 5 mHz convex transducer for the abdominal aorta, by an expert sonographer and images will be then reviewed offline by an expert vascular surgeon blinded to patients clinical status. Ultrasonography of the right and left carotid arteries will be performed in the supine position with the head turned 45° away from the side being imaged. CIMT will be defined as the mean distance from the leading edge of the lumen-intima interface to the leading edge of the media-adventitia interface of the far wall, approximately 10 mm distal to the common carotid artery. CIMT will be calculated by the average of three measurements performed at 0.2 mm intervals.

The abdominal aortic diameter will be measured at maximum systolic expansion (Ds) and minimum diastolic expansion (Dd) at the mid-point between renal arteries origin and iliac carrefour. Aortic strain (S) will be calculated using the formula (S = (Ds-Dd)/Dd). Pressure strain elastic modulus (Ep) will be calculated from S using the formula (Ep=(Ps-Pd)/S; Ps= aortic systolic pressure; Pd= aortic diastolic pressure). Pressure strain normalized by diastolic pressure (Ep*), will be calculated using the formula (Ep* = Ep/Pd). While S is the mean strain of the aortic wall, Ep and Ep* are the mean stiffness of the aorta. To measure brachial artery flow-mediated dilation (FMD), a pneumatic cuff will be placed on the right forearm, 2 cm above the antecubital fossa and inflated to a suprasystolic level (300 mmHg) for 5 minutes. A continuous Doppler velocity assessment will be obtained simultaneously, and data will be collected using the lowest insonation angle (between 30° and 60°). Brachial artery diameters, peak systolic velocity (PSV) and end diastolic velocity (EDV) will be measured immediately after and 2 minutes after the cuff release and then compared to basal values taken immediately before the inflation. The maximum diameter recorded following reactive hyperemia will be reported as a percentage change of resting diameter (FMD = peak diameter - baseline diameter/baseline diameter).

Anthropometric variables Height will be measured to the nearest 0.1 cm using a Harpenden stadiometer, and body weight to the nearest 0.1 kg using a manual weighing scale. Body mass index (BMI) will be calculated as body weight divided by squared height (kg/m2). Waist circumference (WC) will be measured at the high point of the iliac crest around the abdomen and was recorded to the nearest 0.1 cm. Hip circumference will be measured over the widest part of the gluteal region. Pubertal stages will be determined by physical examination, using the criteria of Marshall and Tanner. Systolic (SBP) and diastolic (DBP) blood pressure will be measured three times at 2-minute intervals using a standard mercury sphygmomanometer with an appropriate cuff size. Mean values will be used for the analysis.

Assessment only in the OB group

Biochemical variables After a 12-h overnight fast, blood samples will be taken for measurement of: glucose (mg/dL), insulin (μUI/mL), total cholesterol (mg/dL), high density lipoprotein-cholesterol (HDL-c, mg/dL), triglycerides (mg/dL), sUA (mg/dL), using standardized methods in the Hospital's Laboratory. Low density lipoprotein-cholesterol (LDL-c) will be calculated by the Friedwald formula. sUA (mg/dL) will be measured by Fossati method reaction using uricase with a Trinder-like endpoint.

OB subjects will also undergo an oral glucose tolerance test (1.75 g of glucose solution per kg, maximum 75 g) and samples will be drawn for the determination of glucose and insulin every 30 min. Insulin-resistance at fasting will be calculated using the formula of homeostasis model assessment (HOMA)-IR. Insulin sensitivity at fasting and during OGTT will be calculated as the formula of the Quantitative Insulin-Sensitivity Check Index (QUICKI) and Matsuda index (ISI).

Determination of interleukins (IL), tumor necrosis factor (TNF)α, plasminogen activator inhibitor-1 (PAI1), adiponectin and plasmatic markers of oxidative stress IL-8, IL-10, IL-6, TNFα, PAI-1, adiponectin, 3-nitrotyrosine, malondialdehyde (MDA), reactive oxygen species (ROS) generation, myeloperoxidase (MPO), reduced glutathione (GSH) and superoxide dismutase (SOD) will be measured using specific kits. NO will be quantified from blood samples by using the Griess reagent.

Mitochondria morphology and function Mitochondria will be isolated from monocytes. Ultrastructural analyses of mitochondria (through transmission electron microscope ZEISS 109) will be performed to assess morphologic mitochondrial changes (mitochondrial swelling, decrease in matrix density, possible difference in the sub-plasmalemmal and intrafibrillar sub-fraction of mitochondria, fission-fusion dynamic mitochondrial propriety, mitophagy). Moreover, mitochondria will be used for in vitro assays of mitochondrial oxygen consumption, complex I activity (NAD+/NADH), transmembrane potential and mitochondrial dynamic proteins expression (fusion and fission ratio through mitofusin 1 and 2 Western blot analysis).

Time course of measurements in the OB group All the evaluations previously described will be performed at baseline and after 6 (T6) and 12 months (T12) of an isocaloric Mediterranean balanced diet plus aerobic training.

Nutritional analysis and interventions A well-trained and experienced clinical paediatric endocrinologist will assess food consumption in all subjects and will administer an isocaloric Mediterranean balanced diet in OB children. To assess food consumption, foods will be divided according to the classic basic food groups by the Italian Institute of Research on Food and Nutrition. Food frequencies questionnaires, validated for a wide range of ages, will be also completed by parents. The nutritional counselling will be performed at baseline and after 6 and 12 months, according to Italian LARN (Livelli di Assunzione di Riferimento di Nutrienti) Guidelines and the Italian food pyramid.

Moreover, obese subjects will undergo an exercise training regimen. Exercise will be conducted daily and will consist of 60 minutes of aerobic physical activity. Parents will record every day, on a specific questionnaire, the training performed.

ELIGIBILITY:
Inclusion Criteria:

* children and adolescents (6-16 years);
* obese (OB) and normal weight (NW, control group) according to the International Obesity Task Force (IOTF) criteria;
* both genders;
* diet naïve.

Exclusion Criteria:

* specific causes of endocrine or genetic obesity;
* type 1 or type 2 diabetes;
* previous heart, respiratory, liver and kidney diseases,
* current or past use of hormonal or interfering therapies (lipid-lowering, hypoglycemic, or antihypertensive treatments).

Ages: 6 Years to 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 100 (Actual)
Dates: Start 2015-01-15 (Actual); Primary Completion 2017-02-08 (Actual); Study Completion 2023-07-21 (Actual)

PRIMARY OUTCOMES:
Early cardiovascular abnormalities in OB patients compared with NW subjects | Baseline: at study entry
  We performed transthoracic echocardiogram to all subjects. Measurements of left ventricle (LV), left atrium diameter (LAD), LA and LV volumes, LV systolic and diastolic function, LV mass and relative wall thickness were obtained and compared between OB and matched NW subjects. A vascular assessment was also performed which included carotid artery intima-media thickness (CIMT), abdominal aortic strain and stiffness and brachial artery flow-mediated dilation (FMD). All these measurements were compared between OB and NW subjects. A sample of 15 individuals has been estimated to be sufficient to demonstrate a difference of 10% in LV diameter with a standard deviation (SD) of 0.44 cm with 90% power and a significance level of 95% in the Student t-test between OB and NW according to published data.

SECONDARY OUTCOMES:
Potential association of cardiovascular abnormalities with insulin resistance (IR) in the OB group | Baseline: at study entry
  In the OB group, after a 12-h overnight fast, blood samples were taken for measurement of glucose and insulin using standardized methods in the Hospital's Laboratory. Obese subjects also underwent an OGTT. Insulin-resistance at fasting was calculated using the formula of homeostasis model assessment (HOMA)-IR. Insulin sensitivity at fasting and during OGTT was calculated as the formula of the Quantitative Insulin-Sensitivity Check Index (QUICKI) and Matsuda index (ISI).
Potential association of cardiovascular abnormalities with serum uric acid (sUA) in the OB group | Baseline: at study entry
  In the OB group, after a 12-h overnight fast, blood samples were taken for measurement of sUA using standardized methods in the Hospital's Laboratory. sUA was measured by Fossati method reaction.
Potential association of cardiovascular abnormalities with metabolic syndrome (MetS) in the OB group | Baseline: at study entry
  MetS was defined by using the modified National Cholesterol Education Program/Adult Treatment Panel III (NCEP-ATP III) criteria. A cohort of 75 obese subjects has been estimated to be sufficient to demonstrate differences among numbers of MetS criteria (0-5 criteria according to NCEP-ATPII classification).
Variations of cardiovascular abnormalities in the OB group after 6 and 12 months of behavioral treatment | After 6 and 12 months of behavioral (diet plus aerobic training) treatment
  OB subjects will perform cardiovascular assessment after 6 and 12 months of isocaloric Mediterranean balanced diet plus aerobic training.
Association of cardiovascular abnormalities with IR in the OB group after 6 and 12 months of behavioral treatment | After 6 and 12 months of behavioral (diet plus aerobic training) treatment
  In the OB group, after 6 and 12 month of behavioral treatment, blood samples were taken for measurement of glucose and insulin. Obese subjects also underwent an OGTT. Insulin-resistance at fasting was calculated using the formula of homeostasis model assessment (HOMA)-IR. Insulin sensitivity at fasting and during OGTT was calculated as the formula of the Quantitative Insulin-Sensitivity Check Index (QUICKI) and Matsuda index (ISI). IR will be correlated with cardiovascular measurements
Association of cardiovascular abnormalities with sUA in the OB group after 6 and 12 months of behavioral treatment | After 6 and 12 months of behavioral (diet plus aerobic training) treatment
  In the OB group, after 6 and 12 month of behavioral treatment, blood samples were taken for measurement of sUA. sUA will be correlated with cardiovascular measurements.
Association of cardiovascular abnormalities with MetS in the OB group after 6 and 12 months of behavioral treatment | After 6 and 12 months of behavioral (diet plus aerobic training) treatment
  In the OB group, after 6 and 12 month of behavioral treatment, the presence of MetS was evaluated. The presence/absence of MetS and the number of MetS criteria were correlated with cardiovascular measurements.
Association between cardiovascular dysfunction and adiponectin, inflammatory and oxidative stress plasmatic markers. | Baseline and after 6 and 12 months of behavioral (diet plus aerobic training) treatment
  In the OB group at all study time points, blood samples will be stored and will be analyzed for: IL-8, IL-10, IL-6, TNFα, PAI-1, adiponectin, 3-nitrotyrosine, MDA, ROS generation, MPO, GSH, SOD and NO. An ultrastructural and functional analysis of mitochondria will be also performed. All these dosages will be correlated with cardiovascular abnormalities.

CONTACTS AND LOCATIONS:
Overall Officials: Flavia Prodam, Prof, Principal Investigator — Division of Pediatrics, Department of Health Sciences, University of Piemonte Orientale, Novara, Italy

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Ebbeling CB, Pawlak DB, Ludwig DS. Childhood obesity: public-health crisis, common sense cure. Lancet. 2002 Aug 10;360(9331):473-82. doi: 10.1016/S0140-6736(02)09678-2. PMID 12241736
- [Background] Guo SS, Wu W, Chumlea WC, Roche AF. Predicting overweight and obesity in adulthood from body mass index values in childhood and adolescence. Am J Clin Nutr. 2002 Sep;76(3):653-8. doi: 10.1093/ajcn/76.3.653. PMID 12198014
- [Background] Freedman DS, Khan LK, Dietz WH, Srinivasan SR, Berenson GS. Relationship of childhood obesity to coronary heart disease risk factors in adulthood: the Bogalusa Heart Study. Pediatrics. 2001 Sep;108(3):712-8. doi: 10.1542/peds.108.3.712. PMID 11533341
- [Background] McGill HC Jr, McMahan CA, Zieske AW, Tracy RE, Malcom GT, Herderick EE, Strong JP. Association of Coronary Heart Disease Risk Factors with microscopic qualities of coronary atherosclerosis in youth. Circulation. 2000 Jul 25;102(4):374-9. doi: 10.1161/01.cir.102.4.374. PMID 10908207
- [Background] Sivanandam S, Sinaiko AR, Jacobs DR Jr, Steffen L, Moran A, Steinberger J. Relation of increase in adiposity to increase in left ventricular mass from childhood to young adulthood. Am J Cardiol. 2006 Aug 1;98(3):411-5. doi: 10.1016/j.amjcard.2006.02.044. Epub 2006 Jun 12. PMID 16860034
- [Background] Chinali M, de Simone G, Roman MJ, Lee ET, Best LG, Howard BV, Devereux RB. Impact of obesity on cardiac geometry and function in a population of adolescents: the Strong Heart Study. J Am Coll Cardiol. 2006 Jun 6;47(11):2267-73. doi: 10.1016/j.jacc.2006.03.004. PMID 16750694
- [Background] Dhuper S, Abdullah RA, Weichbrod L, Mahdi E, Cohen HW. Association of obesity and hypertension with left ventricular geometry and function in children and adolescents. Obesity (Silver Spring). 2011 Jan;19(1):128-33. doi: 10.1038/oby.2010.134. Epub 2010 Jun 17. PMID 20559301
- [Background] Sharpe JA, Naylor LH, Jones TW, Davis EA, O'Driscoll G, Ramsay JM, Green DJ. Impact of obesity on diastolic function in subjects < or = 16 years of age. Am J Cardiol. 2006 Sep 1;98(5):691-3. doi: 10.1016/j.amjcard.2006.03.052. Epub 2006 Jul 7. PMID 16923463
- [Background] Mahfouz RA, Dewedar A, Abdelmoneim A, Hossien EM. Aortic and pulmonary artery stiffness and cardiac function in children at risk for obesity. Echocardiography. 2012 Sep;29(8):984-90. doi: 10.1111/j.1540-8175.2012.01736.x. Epub 2012 Jun 14. PMID 22694671
- [Background] Cote AT, Harris KC, Panagiotopoulos C, Sandor GG, Devlin AM. Childhood obesity and cardiovascular dysfunction. J Am Coll Cardiol. 2013 Oct 8;62(15):1309-19. doi: 10.1016/j.jacc.2013.07.042. Epub 2013 Aug 14. PMID 23954339
- [Background] Meyer AA, Kundt G, Steiner M, Schuff-Werner P, Kienast W. Impaired flow-mediated vasodilation, carotid artery intima-media thickening, and elevated endothelial plasma markers in obese children: the impact of cardiovascular risk factors. Pediatrics. 2006 May;117(5):1560-7. doi: 10.1542/peds.2005-2140. PMID 16651309
- [Background] Soltani Z, Rasheed K, Kapusta DR, Reisin E. Potential role of uric acid in metabolic syndrome, hypertension, kidney injury, and cardiovascular diseases: is it time for reappraisal? Curr Hypertens Rep. 2013 Jun;15(3):175-81. doi: 10.1007/s11906-013-0344-5. PMID 23588856
- [Background] Cole TJ, Lobstein T. Extended international (IOTF) body mass index cut-offs for thinness, overweight and obesity. Pediatr Obes. 2012 Aug;7(4):284-94. doi: 10.1111/j.2047-6310.2012.00064.x. Epub 2012 Jun 19. PMID 22715120
- [Background] Cruz ML, Goran MI. The metabolic syndrome in children and adolescents. Curr Diab Rep. 2004 Feb;4(1):53-62. doi: 10.1007/s11892-004-0012-x. PMID 14764281
- [Background] Alpert MA. Obesity cardiomyopathy: pathophysiology and evolution of the clinical syndrome. Am J Med Sci. 2001 Apr;321(4):225-36. doi: 10.1097/00000441-200104000-00003. PMID 11307864
- [Background] Reinehr T, Kiess W, de Sousa G, Stoffel-Wagner B, Wunsch R. Intima media thickness in childhood obesity: relations to inflammatory marker, glucose metabolism, and blood pressure. Metabolism. 2006 Jan;55(1):113-8. doi: 10.1016/j.metabol.2005.07.016. PMID 16324929
- [Background] Ford ES, Li C, Cook S, Choi HK. Serum concentrations of uric acid and the metabolic syndrome among US children and adolescents. Circulation. 2007 May 15;115(19):2526-32. doi: 10.1161/CIRCULATIONAHA.106.657627. Epub 2007 Apr 30. PMID 17470699
- [Background] Sun D, Li S, Zhang X, Fernandez C, Chen W, Srinivasan SR, Berenson GS. Uric acid is associated with metabolic syndrome in children and adults in a community: the Bogalusa Heart Study. PLoS One. 2014 Oct 24;9(10):e89696. doi: 10.1371/journal.pone.0089696. eCollection 2014. PMID 25343690
- [Background] Mangge H, Zelzer S, Puerstner P, Schnedl WJ, Reeves G, Postolache TT, Weghuber D. Uric acid best predicts metabolically unhealthy obesity with increased cardiovascular risk in youth and adults. Obesity (Silver Spring). 2013 Jan;21(1):E71-7. doi: 10.1002/oby.20061. Epub 2013 Jan 29. PMID 23401248
- [Background] Krishnan E, Hariri A, Dabbous O, Pandya BJ. Hyperuricemia and the echocardiographic measures of myocardial dysfunction. Congest Heart Fail. 2012 May-Jun;18(3):138-43. doi: 10.1111/j.1751-7133.2011.00259.x. Epub 2011 Oct 31. PMID 22587743
- [Background] Valle M, Martos R, Canete MD, Valle R, van Donkelaar EL, Bermudo F, Canete R. Association of serum uric acid levels to inflammation biomarkers and endothelial dysfunction in obese prepubertal children. Pediatr Diabetes. 2015 Sep;16(6):441-7. doi: 10.1111/pedi.12199. Epub 2014 Aug 18. PMID 25131560
- [Background] Van Gaal LF, Mertens IL, De Block CE. Mechanisms linking obesity with cardiovascular disease. Nature. 2006 Dec 14;444(7121):875-80. doi: 10.1038/nature05487. PMID 17167476
- [Background] Kershaw EE, Flier JS. Adipose tissue as an endocrine organ. J Clin Endocrinol Metab. 2004 Jun;89(6):2548-56. doi: 10.1210/jc.2004-0395. PMID 15181022
- [Background] Beltowski J, Jamroz-Wisniewska A, Widomska S. Adiponectin and its role in cardiovascular diseases. Cardiovasc Hematol Disord Drug Targets. 2008 Mar;8(1):7-46. doi: 10.2174/187152908783884920. PMID 18336252
- [Background] Ouchi N, Walsh K. Adiponectin as an anti-inflammatory factor. Clin Chim Acta. 2007 May 1;380(1-2):24-30. doi: 10.1016/j.cca.2007.01.026. Epub 2007 Feb 2. PMID 17343838
- [Background] Barseghian A, Gawande D, Bajaj M. Adiponectin and vulnerable atherosclerotic plaques. J Am Coll Cardiol. 2011 Feb 15;57(7):761-70. doi: 10.1016/j.jacc.2010.11.011. PMID 21310310